CLINICAL TRIAL: NCT02987049
Title: Intensive Cardiac Rehabilitation (ICR) With the Pritikin Program: Tolerability and Effectiveness
Brief Title: Intensive Cardiac Rehabilitation (ICR): Tolerability and Effectiveness
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201611030
Record Dates: First submitted 2016-11-16; First posted 2016-12-08 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Disease
Keywords: heart disease, cardiac rehabilitation
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained and the serum or plasma will be stored for future quantification of inflammatory cytokines and other factors related to cardiovascular disease risk.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICR (Intensive Cardiac Rehab): The Intensive Cardiac Rehabilitation (ICR) group will follow their physician-prescribed series of supervised exercise sessions and educational sessions in a cardiac rehab facility. The education component includes a series of Pritikin videos, nutrition workshops and cooking classes led by a registered dietitian, one-on-one dietary consultation with a registered dietitian, and a Pritikin notebook. The intervention for this study is comprised of 24 exercise sessions plus 24 educational sessions in 24 visits.
- CR (conventional Cardiac Rehab): The conventional Cardiac Rehabilitation (CR) group will follow their physician-prescribed series of supervised exercise sessions in the same cardiac rehab facility as the ICR group. The intervention for this study is comprised of 24 exercise sessions during 24 visits.

SUMMARY:
The purpose of this study is to fill in the gaps in knowledge on the tolerability and effectiveness of an outpatient, Pritikin-based Intensive Cardiac Rehabilitation (ICR) program on traditional cardiovascular risk factors, exercise performance, and patient well-being (as assessed by questionnaires), as well as to monitor subsequent clinical events. The hypothesis is that patients in the Intensive Cardiac Rehabilitation (ICR) group will have greater improvements in several cardiovascular disease risk factors than patients in the conventional Cardiac Rehabilitation (CR) group at the end of 24 sessions.

DETAILED DESCRIPTION:
BACKGROUND: Conventional Cardiac Rehabilitation (CR) involves a 36-session supervised and monitored exercise treatment program in a cardiac rehabilitation facility for patients with an approved cardiac diagnosis, such as chronic angina, recent myocardial infarction (heart attack), cardiac surgery, or recent percutaneous coronary intervention. The exercise sessions generally are one hour each and the treatment period is typically over 12 weeks. Intensive Cardiac Rehabilitation (ICR) includes the 36-session exercise intervention plus 36 one-hour educational sessions on the Pritikin program. These education sessions include one-on-one dietary consultation with a registered dietitian, nutrition workshops and cooking classes led by a registered dietitian, a series of Pritikin videos, and a notebook of Pritikin handouts on various topics, including reading nutrition labels, how to prepare heart-healthy meals, mindfulness, smoking cessation, and the process of atherosclerosis.

Nathan Pritikin started the Pritikin program in the 1970s with the aim of decreasing recurrent cardiovascular disease (CVD) events in humans. The three pillars of the Pritikin lifestyle program are a healthy diet, exercise, and mindfulness. The Pritikin diet emphasizes unprocessed foods that are high in fiber, low in calorie density, and very low in sodium, saturated fat, and cholesterol. Mindfulness includes behavior modification therapies such as smoking cessation and stress management. Since the 1970s, there have been more than 100 publications in scientific, peer-reviewed journals demonstrating the efficacy of this program on improving many traditional cardiac risk factors and biomarkers of cardiac health, as well as preventing and treating CVD. In addition, a low-fat, high fiber diet combined with exercise has been shown to improve markers of nitric oxide bioavailability and fasting insulin concentrations.

Most of these results, however, were derived from studies of patients domiciled at a Pritikin wellness center. Relatively recently, the Pritikin program was approved as a form of ICR in an outpatient setting. The BJC/Washington University School of Medicine Cardiac Rehab program at the Heart Care Institute was the first Cardiac Rehab program in the world to offer an outpatient Pritikin ICR program. Currently, Medicare and some (but not all) third-party insurance companies pay for ICR. Thus, many patients under the age of 65 years are not afforded the potential benefits of ICR.

SPECIFIC AIM: The purpose of this study is to fill in the gaps in knowledge on the tolerability and effectiveness of an outpatient, Pritikin-based ICR program on traditional cardiovascular risk factors, exercise performance, and patient well-being (as assessed by questionnaires), as well as to monitor subsequent clinical events in this outpatient population.

HYPOTHESIS: The hypothesis is that patients in the Intensive Cardiac Rehabilitation (ICR) group will have greater improvements in several cardiovascular risk factors than patients in the conventional Cardiac Rehab (CR) group at the end of 24 sessions.

FUTURE DIRECTIONS: If the results of this study are favorable, then there are several implications for clinical practice. 1) Evidence of the effectiveness and tolerability of outpatient ICR should encourage expanded coverage of ICR so that more cardiac patients may benefit from this treatment in the future. 2) Demonstration of any trends in improvement of outcomes would support the need for a multi-center trial to define the degree to which ICR can help patients and decrease health care-related costs. These questions would be explored in future R34 grants and Patient-Centered Outcomes Research Institute (PCORI) grants.

STUDY OVERVIEW: This is a 2-year, non-randomized study in which the Intensive Cardiac Rehab (ICR) and conventional Cardiac Rehab (CR) treatment programs are already being conducted as part of routine clinical care in a cardiac rehabilitation facility. Many of the assessments to be conducted and the outcome measures of this study are being obtained as part of the existing cardiac rehab programs. Assignment to the ICR or CR group will be according to the referring physician's recommendation and insurance coverage and will occur before study enrollment. The research portion is obtaining permission to include the participants' phenotypic and outcome data in the research study database and analyzing the information in a systematic manner to answer study questions regarding the tolerability and effectiveness of the ICR program. Participants also will be asked to complete additional assessments and questionnaires that are for research purposes only.

ELIGIBILITY:
Inclusion Criteria:

* individuals with a cardiac diagnosis or procedure who are referred to the BJC HealthCare / Washington University School of Medicine Cardiac Rehab program at the Heart Care Institute in St. Louis, Missouri
* individuals who are ambulatory

Exclusion Criteria:

* individuals with other significant medical conditions that preclude exercise or that would interfere with the assessments involved in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients who are at least 18 years of age and are referred to the BJC/Washington University School of Medicine Cardiac Rehab program at the Heart Care Institute in St. Louis, MO will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Baseline and Vist 24, which occurs between 8 and 12 weeks
  BMI will be computed from measured height and weight

SECONDARY OUTCOMES:
Dietary Intake | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Diet will be assessed using the Rate Your Plate questionnaire
Body Composition | Baseline and Vist 24, which occurs between 8 and 12 weeks
  % body fat, fat mass (kg), and fat-free mass (FFM) will be assessed by bioelectrical impedance analysis

OTHER OUTCOMES:
Hand Grip Strength | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Quantified with a Jamar Plus hand dynamometer
Short Physical Performance Battery (SPBB) | Baseline and Vist 24, which occurs between 8 and 12 weeks
  3 tests: 4m walk, balance, chair rise
Serum Lipid Concentrations | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides
Hemoglobin A1c | Baseline and Vist 24, which occurs between 8 and 12 weeks
  quantified in whole blood
Resting Blood Pressure | Baseline and Vist 24, which occurs between 8 and 12 weeks
  systolic BP and diastolic BP (mmHg)
Resting Heart Rate | Baseline and Vist 24, which occurs between 8 and 12 weeks
  bpm
Duke Activity Status Index (DASI) Questionnaire | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Self-reported physical activity assessment
Dartmouth Coop General Health Questionnaire | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Self-reported general health
Cardiac Self-Efficacy Questionnaire | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Sullivan CSE
Patient Health Questionnaire-9 (PHQ-9) | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Depression assessment
6-Minute Walk | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Distance walked in 6 minutes
Arterial Function | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Endothelial vasodilator function (i.e., arterial function) will be assessed using an EndoPat device
Medication Changes | Baseline and Vist 24, which occurs between 8 and 12 weeks
  Medication changes from Baseline to Visit 24

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Peterson, MD, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided
The current plan is that individual participant data will be shared with investigators on the research team only.

REFERENCES:
- [Background] Martin W. Nathan Pritikin and atheroma. Med Hypotheses. 1991 Nov;36(3):181-2. doi: 10.1016/0306-9877(91)90125-i. No abstract available. PMID 1787805
- [Background] Rosenthal MB, Barnard RJ, Rose DP, Inkeles S, Hall J, Pritikin N. Effects of a high-complex-carbohydrate, low-fat, low-cholesterol diet on levels of serum lipids and estradiol. Am J Med. 1985 Jan;78(1):23-7. doi: 10.1016/0002-9343(85)90456-5. PMID 3966484
- [Background] Roberts CK, Vaziri ND, Barnard RJ. Effect of diet and exercise intervention on blood pressure, insulin, oxidative stress, and nitric oxide availability. Circulation. 2002 Nov 12;106(20):2530-2. doi: 10.1161/01.cir.0000040584.91836.0d. PMID 12427646